CLINICAL TRIAL: NCT03194425
Title: Pelvic Floor EMG Monitoring as Tool to Improve Patient Selection and Outcome - Standardization of Lead Placement for Sacral Neuromodulation.
Brief Title: Standardization of Lead Placement for Sacral Neuromodulation. Part 1
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universiteit Antwerpen (Other)
Collaborators: Leiden University Medical Center (Other)
Responsible Party: Principal Investigator, Donald Vaganée, Principal Investigator, Universiteit Antwerpen
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: B300201523497 Part 1
Record Dates: First submitted 2017-05-10; First posted 2017-06-21 (Actual); Last update posted 2019-10-15 (Actual); Status verified 2019-10

CONDITIONS: Overactive Bladder; Non Obstructive Urinary Retention
Keywords: Sacral neuromodulation; Electromyography; Pelvic floor
MeSH Terms: conditions — Urinary Bladder, Overactive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OAB (Experimental): Patients with overactive bladder on sacral neuromodulation.
  Interventions: Diagnostic Test: Pelvic floor EMG
- NOUR (Experimental): Patients with non-obstructive urinary retention on sacral neuromodulation.
  Interventions: Diagnostic Test: Pelvic floor EMG

INTERVENTIONS:
Diagnostic Test: Pelvic floor EMG — Define pelvic floor EMG template measured by probe

SUMMARY:
Retrospective case-control study.

A substantial number of patients do not respond favourably to sacral neurostimulation (SNS) although clinically, they appear to have the same lower urinary tract dysfunction characteristics as the ones with good responses. This may be due to methodological issues (lead position) or patient selection. The purpose of this study is to improve and standardize lead position, in order to increase the patient response to test stimulation and to SNS treatment, and to decrease adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged ≥18 years and competent to provide consent
2. Minimum 3 months of self-reported OAB symptoms or self-reported obstructive LUTS in addition to confirmed non-obstructive urinary retention on UDO
3. Failed, or are not a candidate for more conservative treatment (i.e., pelvic floor training, biofeedback, behavioral modification, oral pharmacotherapy)
4. Willing to discontinue OAB medications for 2 weeks prior to the implant and for the entire study period
5. Able to thoroughly fill in all questionnaires, voiding diaries and office visits for device programming and clinical evaluations before the TLP, 3 weeks after TLP and 6 weeks, 6 months and 1 year after implantation of definitive IPG.

Exclusion Criteria:

1. Current of prior evidence of primary stress incontinence or mixed incontinence where the stress component overrides the urgency component
2. Any neurological condition that may interfere with normal bladder function, including stroke, multiple sclerosis, Parkinson's disease, clinically significant peripheral neuropathy, or spinal cord injury (e.g., paraplegia)
3. Urinary tract mechanical obstruction including but not limited to Benign Prostatic Hyperplasia (BPH)
4. Treatment of bladder or pelvic floor dysfunction with botulinum toxin (Botox ®) or surgery in past 12 months
5. Unable to toilet self and have and maintain good personal hygiene
6. Unable to provide clear, thoughtful responses to questions and questionnaires
7. Urinary tract, bladder or vaginal infection or inflammation
8. Hematuria, and absence of an elaborate diagnostic work-up
9. Severe or uncontrolled diabetes (A1C > 8, documented in the last 3 months) or diabetes with peripheral nerve involvement
10. Allergy to local anesthetic or adhesives
11. Bleeding disorder or on an anticoagulant that cannot be stopped for 3 days before the implant
12. Pregnant, lactating, planning to become pregnant, given birth in the past 12 months, or female of child-bearing potential and not practicing a medically-approved method of birth control
13. Skin lesions or compromised skin at the implant or stimulation site
14. Use of investigational drug or device therapy or participation in any study involving or impacting gynecologic, urinary or renal function within past 4 weeks
15. Passive implants (e.g., prostheses) are allowed, but no implanted metal should be at the Neurostimulator implant site
16. Knowledge of planned MRIs, diathermy, or high output ultrasonic exposure
17. Presence of a documented condition or abnormality that could compromise the safety of the patient
18. Any psychiatric or personality disorder at the discretion of the study physician
19. Interstitial cystitis or bladder pain syndrome as defined by the EAU guidelines
20. Life expectancy of less than 1 year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-09-01 (Actual); Primary Completion 2022-08 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
EMG activity of pelvic floor muscles in OAB patients and NOUR patients already on SNM | 1 day
  Latency and amplitude of pelvic floor measured by EMG probe

CONTACTS AND LOCATIONS:
Overall Officials: Stefan De Wachter, MD PhD FEBU, Study Director — University Hospital, Antwerp; Donald Vaganée, Principal Investigator — University Hospital, Antwerp
Locations (1):
- Antwerp University Hospital, Edegem, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: No